CLINICAL TRIAL: NCT00152659
Title: Developing Functional and Structural Criteria for Cortical Resections
Brief Title: Developing Criteria for Cortical Resections
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 9538
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Epilepsy; Tumor
Keywords: Epilepsy; Tumor; Surgery; Brain
MeSH Terms: conditions — Epilepsy; Neoplasms | interventions — Histocompatibility Testing; Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Tissue sample (procedure/screening) — Tissue sampling

SUMMARY:
The purpose of this study is to study how disease processes like tumors or epilepsy spread in the brain.

DETAILED DESCRIPTION:
The purpose of this study is to study how disease processes like tumors or epilepsy spread in the brain. During surgery small pieces of abnormal (unusual) brain tissue may be removed. We analyze these specimens using more advanced microscopic and electrophysiologic techniques than are usually applied to such tissue specimens. In addition, some tissues can be maintained in laboratory conditions to allow analysis over the longer term. No extra brain tissue is taken to perform these studies. The tissue analysis is performed by the research team and are compared to the routine (normal) electrical recordings that are taken during this type of brain surgery. Currently there are no instructions telling a doctor how much brain tissue should be cut out to prevent the spread of tumors or epilepsy. We are hoping that the results of this study help us to better know how much brain tissue needs to be removed to prevent the spread of tumors or epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidates with epilepsy or brain tumor(s)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical candidates with epilepsy or brain tumor(s)
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 1998-09-01 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
measure electrical activity in tissue sample | at tissue aremoval time

CONTACTS AND LOCATIONS:
Overall Officials: Wim van Drongelen, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Hospitals, The University of Chicago Comer Children's Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Ramirez J-M, Koch H, Pena F, Drongelen W van, Tryba AK, Parkis MA, Loweth JA, Hecox KE, Kohrman MH, Frim DM, Chico MS, Marcuccilli CJ (2003) - In vitro electrophysiological differences between least and most abnormal tissue obtained from pediatric patients with intractable epilepsy. Epilepsia 44, Suppl 9: 245-246
- [Background] Marcuccilli CJ, Koch H, Pena F, Drongelen W van, Tryba AK, Parkis MA, Hecox KE, Kohrman MH, Frim DM, OConnor SE, Chico MS, Ramirez J-M (2003) - Rational pharmacotherapy: relationship between in vitro electrophysiology and clinical measures. Epilepsia 44, Suppl 9: 244-245
- [Background] Drongelen W van, Koch H, Marcuccilli CJ, Viemari J, Tryba AKH, Loweth JA, Ramirez J-M, Elsen F (2004) - Persistent sodium current plays a critical role in the generation of slow oscillations in vitro neocortex brain slices of mice and humans. Abstract Soc Neuroscience
- [Background] Drongelen W van, Doren EL, Koch H, Marcuccilli CJ, Ramirez J-M, Elsen FP (2005) - Characterization of the persistent sodium current in neocortical networks of mice and humans. Abstract Washington DC: Society for Neuroscience